CLINICAL TRIAL: NCT00337493
Title: A Study to Investigate the Impact of Pharmacogenetics on CellCept Use, in Patients Participating in a Study in Renal Transplantation
Brief Title: Pharmacogenetic Study of CellCept (Mycophenolate Mofetil) in Kidney Transplant Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19199
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Cyclosporine; Tacrolimus

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: mycophenolate mofetil [CellCept]; Drug: Cyclosporine or tacrolimus
- 2 (Experimental)
  Interventions: Drug: mycophenolate mofetil [CellCept]; Drug: Cyclosporine or tacrolimus
- 3 (Experimental)
  Interventions: Drug: mycophenolate mofetil [CellCept]; Drug: Cyclosporine or tacrolimus

INTERVENTIONS:
Drug: mycophenolate mofetil [CellCept] — Concentration-controlled
  Arms: 1; 2
Drug: mycophenolate mofetil [CellCept] — 1g po bid
  Arms: 3
Drug: Cyclosporine or tacrolimus — Reduced
  Arms: 1
Drug: Cyclosporine or tacrolimus — Standard, as prescribed
  Arms: 2; 3

SUMMARY:
This study will determine which, if any, allelic variants of mycophenolic acid (MPA) metabolizing enzymes, drug transporters and drug targets are associated with the observed variation in pharmacokinetic and pharmacodynamic outcomes observed with CellCept usage. Patients participating in study ML17225 will be eligible for this pharmacogenetic investigation, and will have one additional blood sample taken during the study. The anticipated time on study treatment in study ML17225 is 1-2 years, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients participating in study ML17225.

Exclusion Criteria:

* N/A.

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Correlation of allelic variants of MPA metabolizing genes, membrane transporter genes and target genes with AUC, transplant rejection, GER and drug side effects. | Throughout study

SECONDARY OUTCOMES:
Viral kinetics | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- United States (20):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - Denver, Colorado
  - Gainesville, Florida
  - Orlando, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Hackensack, New Jersey
  - Livingston, New Jersey
  - Buffalo, New York
  - Chapel Hill, North Carolina
  - Fargo, North Dakota
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Madison, Wisconsin